CLINICAL TRIAL: NCT05319665
Title: "connEcted Caesarean Section": Creating a Virtual Link Between MOthers and Their infanTs to ImprOve Maternal Childbirth experieNce: a PILOT Trial (E-motion-pilot)
Brief Title: "Connected Caesarean Section": Creating a Virtual Link Between Mothers and Their Infants to Improve Maternal Childbirth Experience: A Pilot Trial
Acronym: e-motion-pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Principal Investigator, Antje Horsch, Associate Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2022-00215
Record Dates: First submitted 2022-03-25; First posted 2022-04-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Post Traumatic Stress Disorder; Childbirth Experience
Keywords: Mother-infant bonding; Birth satisfaction; HMD; Virtual reality; Caesarean section
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Smart Glasses

STUDY DESIGN:
Intervention Model Description: The study will consist of two phases. During the first phase, the participants will be the control group and will have the standard-of-care. During the second phase, the participants will be the interventional group and will have a head-mounted display airing a live video of their newborn filmed by a 2D 360° camera to enable a visual and auditory contact.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will have the standard-of-care treatment.
- Interventional (Experimental): The interventional group will have a head-mounted display whilst still in the operating theatre airing a live video of their newborn filmed by a 2D 360° camera to enable a visual and auditory contact.
  Interventions: Device: Head-mounted display

INTERVENTIONS:
Device: Head-mounted display — The intervention is a visual and auditory contact via a head-mounted display (HMD) worn by the mother airing a live video of her newborn filmed by a 2D 360° camera during and after a caesarean section. The HMD will be worn by the new mother from the moment that her newborn is moved to an adjacent room to receive the initial care until the moment when they can be reunited again. The camera will be placed in the adjacent room where the newborn, the mother's partner and a midwife will be. The camera will film the newborn and transmit the live images and the sound to the HMD worn by the mother. The mother will be able to see and hear what happens in the next room and change her angle of view by moving her head from one side to another.
  Arms: Interventional

SUMMARY:
One third of mothers rate their childbirth as traumatic. The prevalence of childbirth-related posttraumatic stress disorder (CB-PTSD) is of 4.7% and the prevalence of childbirth-related posttraumatic stress symptoms (CB-PTSS) of 12.3%. Skin-to-skin contact is a protective factor against CB-PTSD. However, during a caesarean section (CS), skin-to-skin contact is not always feasible and mothers and infants are often separated. In those cases, there is no validated and available solution to substitute this unique protective factor. Based on the results observed in studies using virtual reality (VR) and head-mounted displays (HMDs) and studies on childbirth experience, we hypothesize that enabling the mother to have a visual and auditory contact with her baby could improve her childbirth experience whilst she and her baby are separated. To facilitate this connection, we will use a 2D 360° camera filming the baby linked securely to a head-mounted device (HMD) that the mother can wear during the end of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years old or older
* Planned or unplanned CS at ≥ 34 weeks gestation
* Gave birth to a healthy baby according to pediatric evaluation (APGAR score ≥ 7 at 5 minutes)
* Gave oral consent followed by a written confirmation of consent
* Skin-to-skin contact is not possible or was prematurely interrupted
* Speaks French well enough to participate in study assessments
* Eligibility confirmed by an independent physician for the intervention group
* Partner gave oral consent to be filmed for the intervention group.

Exclusion Criteria:

* Has an established intellectual disability or psychotic illness
* Has photosensitive epilepsy
* Caesarean section under general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Childbirth Experience Questionnaire 2 (CEQ-2) | 1 week after the birth
  Standardised questionnaire of childbirth experience. This self-reported questionnaire measures the maternal childbirth experience with four different subscales: own capacity, perceived safety, professional support and participation. There are 19 items rated on a 4 point Likert scale ranging from 1=totally disagree to 4=totally agree and 3 items rated on a VAS from 1 to 100. Rating of negatively worded statements are reversed. Higher scores indicates a better childbirth experience. The minimum value is 1 and the maximum is 4 points.

SECONDARY OUTCOMES:
Perceived Pain Item | During the caesarean section
  Evaluation of experienced pain using the Pain Item during the caesarean section.
  A visual analogue scale from 0 to 10 will be shown to the participant. She will be asked to evaluate her pain level on that scale. 0 means no pain at all, 10 is the worst pain imaginable.
Perceived Stress Item | At the end of the caesarean section
  Evaluation of experienced the stress using the Stress Item. A visual analogue scale from 0 to 10 will be shown to the participant. She will be asked to evaluate her stess level on that scale. 0 means no stress at all, 10 is the worst stress imaginable.
Perceived Pain Item | At the end of the caesarean section
  Evaluation of experienced pain using the Pain Item. A visual analogue scale from 0 to 10 will be shown to the participant. She will be asked to evaluate her pain level on that scale. 0 means no pain at all, 10 is the worst pain imaginable.
Satisfaction of the intervention | 1 week after the caesarean section
  For the interventional group, their satisfaction of the intervention will be assessed.
  12 questions will be asked to the participants of the interventional group on their global satisfaction of the intervention, the utility of the intervention, the comfort of the HMD, the quality of the images, sound and camera-HMD connection, advantages and disadvantages of the HMD. 3 questions will be evaluated on a 5-point Likert-scale. 4 questions will require a yes-no answer and 5 questions will be open questions.
  This questionnaire is used as a qualitative questionnaire.
Maternal symptoms of anxiety or depression | 1 week after the caesarean section
  Hospital Anxiety and Depression Scale (HADS-A and HADS-D) This self-reported questionnaire measures the severity of anxiety and depression symptoms during the week before replying to the questions. There are two subscales; anxiety and depression. Each of them consists of seven items scored on a four point Likert scale (0= never, 3=most of the time). Higher score reflects greater severity. The minimum value is 0 and the maximum is 42 points.
Mother-infant bonding | 1 week after the caesarean section
  Mother-Infant Bonding Scale (MIBS) This eight points self-reported questionnaire assesses the mother's feelings towards her newborn in the first week after birth. The eights items are statements describing an emotional response and are rated on a four point Likert scale (0=very much, 3=not at all). Higher score denote worse bonding. The minimum value is 0 and the maximum is 24 points.
Satisfaction of the birth | 1 week after the caesarean section
  Birth Satisfaction Scale-Revised (BSS-R) The BSS-R is a 10-item self-reported questionnaire assessing the perceptions of the birth in order to determine women's satisfaction of their birth experience. It consists of one higher-order factor, experience of childbearing, containing three lower-order factors: quality of care provision, women's personal attributes and stress experienced during labor. The items are evaluated on a Likert-type scale that requests participants to rate their level of agreement with each item (1=strongly disagree, 5=strongly agree). Four of the items are reverse-coded. Higher score denotes a worse satisfaction of the birth. The minimum value is 10 and the maximum is 50 points.
Maternal symptoms of anxiety or depression | 1 month after the caesarean section
  Hospital Anxiety and Depression Scale (HADS-A and HADS-D) This self-reported questionnaire measures the severity of anxiety and depression symptoms during the week before replying to the questions. There are two subscales; anxiety and depression. Each of them consists of seven items scored on a four point Likert scale (0= never, 3=most of the time). Higher score reflects greater severity. The minimum value is 0 and the maximum is 42 points.
Maternal symptoms of PTSD | 1 month after the caesarean section
  City Birth Trauma Scale (CityBiTS) (CityBiTS). The City Birth Trauma Scale is a 29-item questionnaire measuring birth-related post-traumatic stress disorder (PTSD) according to DSM-5 criteria of (A) stressor criteria, (B) symptoms of re-experiencing, (C) avoidance, (D) negative cognitions and mood, (E) hyperarousal, (F) duration of symptoms, (E) signification distress or impairment and (F) exclusion criteria or other causes. Items are evaluated with yes/no/maybe or by frequency of the symptoms. A higher score indicates a higher level of PTSD symptoms. The minimum value is 0 and the maximum is 78 points.

OTHER OUTCOMES:
Evolution of the haemodynamic parameters during the caesarean section | During the caesarean section
  The investigators will monitor the haemodynamic parameters during the caesarean section.
  anesthesia, use of medication, Perceived Pain Item
Presence of perioperative shivers during the caesarean section | During the caesarean section
  The investigators will assess if there is a presence of perioperative shivers or not during the caesarean section.
Presence of nausea related to the surgery or the anesthesia during the caesarean section. | During the caesarean section
  The investigators will assess if there is a presence of nausea or not during the caesarean section.
Use of medication during the caesarean section. | During the caesarean section
  The investigators will monitor the use of medication during the caesarean section.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Antje Horsch, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Corbaz F, Boussac E, Lepigeon K, Gomes Dias D, Marcadent S, Desseauve D, Horsch A. 'connEcted caesarean section': creating a virtual link between MOthers and their infanTs to ImprOve maternal childbirth experieNce - study protocol for a PILOT trial (e-motion-pilot). BMJ Open. 2023 Jun 7;13(6):e065830. doi: 10.1136/bmjopen-2022-065830. PMID 37286319